CLINICAL TRIAL: NCT00995735
Title: IMTN Study- International Prospective Multicenter Trial on Clinical NOTES
Acronym: IMTN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IMTN NOTES Research Group (Other)
Responsible Party: Ricardo Zorron, Professor and Chairman, MD, PhD, Brazilian College of Surgeons CBC
Other Study IDs: 0209.0.314.000-08
Record Dates: First submitted 2009-10-14; First posted 2009-10-15 (Estimated); Last update posted 2009-10-15 (Estimated); Status verified 2009-10

CONDITIONS: Gastrointestinal Surgery; Natural Orifice Surgery
Keywords: NOTES; Natural Orifice Translumenal Endoscopic surgery; Cholecystectomy; Appendectomy; Endoscopy; Laparoscopy; Minimally invasive surgery; clinical trials
MeSH Terms: interventions — Cholecystectomy; Appendectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Transgastric: Patients submitted to Transgastric NOTES surgery
  Interventions: Procedure: Cholecystectomy; Procedure: Appendectomy
- Transvaginal: Patients submitted to Transvaginal surgery
  Interventions: Procedure: Cholecystectomy; Procedure: Appendectomy

INTERVENTIONS:
Procedure: Cholecystectomy — Cholecystectomy performed either by entering the stomach wall with the endoscope, or through a posterior vaginal opening.
Procedure: Appendectomy — Appendectomy performed either by entering the stomach wall with the endoscope, or through a posterior vaginal opening.

SUMMARY:
Objectives: Since 2007, natural orifice surgery evolved from theory and animal research to clinical applications, but is still limited in the literature to small casuistic reports. A preliminary prospective evaluation of postoperative results of the early casuistic of Natural orifice Surgery for many indications may show advantages and disadvantages of the methods. The IMTN Multicenter Trial for Clinical NOTES was and early results are described.

ELIGIBILITY:
Inclusion Criteria:

* Patients submitted to elective surgery

Exclusion Criteria:

* emergency surgery High ASA risk patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients submitted to Natural Orifice Surgery with local IRB aproval for human trials.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2007-06; Primary Completion 2009-08 (Actual); Study Completion 2009-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Zorron, Principal Investigator — Brazilian College of Surgeons CBC; Chisunnami Palanivelu, Study Director — Indian Society of Laparoscopic Surgery; Manuel Galvao, Study Director — Society of Brazilian Digestive Endoscopy SOBED; Almino Ramos, Study Director — Brazilian College of Surgeons CBC
Locations (1):
- Hospital Municipal Lourenco Jorge, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Background] Zorron R, Maggioni LC, Pombo L, Oliveira AL, Carvalho GL, Filgueiras M. NOTES transvaginal cholecystectomy: preliminary clinical application. Surg Endosc. 2008 Feb;22(2):542-7. doi: 10.1007/s00464-007-9646-5. Epub 2007 Nov 20. PMID 18027043